CLINICAL TRIAL: NCT01960426
Title: A Randomized Evaluation of Health Costs and Resource Utilization Comparing Testing-Based Therapy to Empiric Dose Intensification for the Management of Inflammatory Bowel Disease.
Brief Title: Evaluation of Health Costs and Resource Utilization
Acronym: Test-NoTest
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment issues
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RP1208
Record Dates: First submitted 2013-09-25; First posted 2013-10-10 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Harvey Bradshaw score; Partial Mayo Clinical Score; Infliximab; Adalimumab
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Adalimumab; Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empiric Dose Intensification (Active Comparator): Intensify treatment with the existing drug
  Interventions: Other: Intensify treatment with the existing drug
- Testing based strategy (Active Comparator): Measurement of drug (Adalimumab/Infliximab) Testing-based strategy for the management of secondary loss of response that is based on drug/ ADA measurement
  Interventions: Other: Measurement of drug (Adalimumab/Infliximab)

INTERVENTIONS:
Other: Measurement of drug (Adalimumab/Infliximab) — Measurement of drug (adalimumab/infliximab) and ADAs in the presence of drug.
  Arms: Testing based strategy
Other: Intensify treatment with the existing drug — Intensify treatment with the existing drug and if this fails empirically switch to another TNF antagonist
  Arms: Empiric Dose Intensification

SUMMARY:
Utilization of health resources in a testing based strategy versus an empiric dose escalation strategy to manage Crohn's disease and Ulcerative Colitis in subjects with loss of response to infliximab or adalimumab.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the utilization of health resources in a testing based strategy versus an empiric dose escalation strategy to manage Crohn's disease and Ulcerative Colitis in subjects with loss of response to infliximab or adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years of age or older who are not receiving azathioprine or 6 mercaptopurine.
* Non-pregnant, non-lactating females, 18 years of age or older.
* Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. [defined as a minimum of one year since the last menstrual period]).
* Documented diagnosis of CD or UC.
* Active disease symptoms at visit 1 defined by: a. CD subjects: HBS ~ 6 UC subjects: PMCS ~ 4.
* Current infliximab therapy (naive to adalimumab) or current adalimumab therapy (naive to infliximab ).
* A minimum of 13 weeks of infliximab or adalimumab treatment prior to visit 1 at the following dose:
* Stable dose of azathioprine, 6 mercaptopurine, methotrexate, and/or 5-aminosalicylates in the 4 weeks prior to visit 1.

Exclusion Criteria:

* Contraindication to the use of either infliximab or adalimumab.
* Current infliximab treatment but not naive to adalimumab or
* Current adalimumab treatment but not naive to infliximab.
* Infliximab dosing prior to visit 1 was not 5 mg/kg at weeks 0, 2 and 6 and then q8w.
* Adalimumab dosing prior to visit 1 was not 160 mg at week 0, 80 mg at week 2, and then 40 mg q2w.
* Received any investigational drug within 30 days prior to visit 1.
* Serious underlying disease other than CD or UC which in the opinion of the investigator may interfere with the subject's ability to participate fully in the study.
* History of alcohol or drug abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
* Stools positive for clostridium difficile.
* Pregnant or lactating women.
* Change in dose of azathioprine, 6 mercaptopurine, methotrexate, and/or 5-aminosalicylates in the 4 weeks prior to visit 1.
* Males 22 years of age or less who are receiving azathioprine or 6 mercaptopurine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
the mean difference in cumulative costs (Visit I to Week 3 1) between the two treatment arms | 31 weeks
  Analysis of costs and outcomes will be made on an intention-to-treat basis

SECONDARY OUTCOMES:
The efficacy of the testing-based strategy compared to empiric dose intensification | 31 weeks
  The proportion of subjects achieving clinical remission

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feagan, MD, Principal Investigator — Robarts Clinical Trials Inc. - Western University
Locations (1):
- Rocky Mountain Gastroenterology Associates, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Velayos FS, Kahn JG, Sandborn WJ, Feagan BG. A test-based strategy is more cost effective than empiric dose escalation for patients with Crohn's disease who lose responsiveness to infliximab. Clin Gastroenterol Hepatol. 2013 Jun;11(6):654-66. doi: 10.1016/j.cgh.2012.12.035. Epub 2013 Jan 26. PMID 23357488
- [Background] Altman DG, Bland JM. Treatment allocation by minimisation. BMJ. 2005 Apr 9;330(7495):843. doi: 10.1136/bmj.330.7495.843. No abstract available. PMID 15817555
- [Background] Hanauer SB, Sandborn WJ, Rutgeerts P, Fedorak RN, Lukas M, MacIntosh D, Panaccione R, Wolf D, Pollack P. Human anti-tumor necrosis factor monoclonal antibody (adalimumab) in Crohn's disease: the CLASSIC-I trial. Gastroenterology. 2006 Feb;130(2):323-33; quiz 591. doi: 10.1053/j.gastro.2005.11.030. PMID 16472588
- [Background] Sandborn WJ, Feagan BG, Stoinov S, Honiball PJ, Rutgeerts P, Mason D, Bloomfield R, Schreiber S; PRECISE 1 Study Investigators. Certolizumab pegol for the treatment of Crohn's disease. N Engl J Med. 2007 Jul 19;357(3):228-38. doi: 10.1056/NEJMoa067594. PMID 17634458